CLINICAL TRIAL: NCT01214785
Title: Assessing the Effect of Improved Rural Sanitation on Diarrhoea and Intestinal Nematode Infections: a Cluster Randomised Controlled Trial in Orissa, India
Brief Title: Cluster Randomised Trial of Improved Sanitation in Rural Orissa, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: WaterAid (Other); Xavier Institute of Management, Bhubaneswar (Other); Bill and Melinda Gates Foundation (Other); International Initiative for Impact Evaluation (Other); Department for International Development, United Kingdom (Other Government); University of California, Davis (Other); Emory University (Other); Asian Institute of Public Health (Other); Kalinga Institute of Industrial Technology (Other)
Responsible Party: Principal Investigator, Thomas Clasen, Dr, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MR03
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Diarrhoea; Soil-transmitted Helminth Infection; Nutritional Status
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sanitation intervention (Active Comparator)
  Interventions: Behavioral: Provision of household latrines
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Provision of household latrines — WaterAid and local NGO partners mobilize householders in target villages to construct and use latrines in accordance with the Government of India's Total Sanitation Campaign.
  Arms: Sanitation intervention

SUMMARY:
The study is a cluster-randomized, controlled trial conducted among 100 villages (including approximately 3500 households and 20,000 people) in Puri district, State of Orissa, India. The study aims to assess the impact of the construction and use of latrines in rural settings on diarrhoeal disease, helminth infections and nutritional status. The study will also report on the cost and cost-effectiveness of the intervention and its impact on lost days at school and work as well as on expenditures on drugs and medical treatment. The study will document how the intervention actually impacts exposure to human excreta along principal transmission pathways by evaluating the impact on (i) faecal contamination of drinking water, (ii) the presence of mechanical vectors (flies) in food preparation areas, and (iii) the presence of faeces in and around participating households and villages. The study will also explore the extent to which different levels of acquisition and use of on-site sanitation among householders impact disease throughout the community.

ELIGIBILITY:
Inclusion Criteria:

Village level:

* Little existing sanitation coverage (<10%)
* WaterAid and implementing partners expects normal scale up
* Stable and reasonably acceptable water supply
* No other WASH interventions planned or anticipated in next 30 months
* Reasonable year-round access by road to permit household visits by surveillance staff

Household level:

* Presence of a child<4 or a pregnant woman
* Consent to participate
* Reside permanently in the village

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Diarrhoea (<5s) | 21 months
  Longitudinal prevalence of diarrhoea (7-day period prevalence) measured repeatedly every 3 months over a 21-month follow-up period. Diarrhoea is defined according to the WHO definition (three of more stools passed in 24 hrs)

SECONDARY OUTCOMES:
Soil-transmitted helminth infection | baseline and endline
  Prevalence of soil-transmitted helminth infection at the end of the follow-up period
Weight-for-age (<5s) | 21 months
  Weight of children <5 is recorded at each diarrhoea surveillance visit (every 3 months over the 21-month follow-up). Weight-for-age Z (WAZ) scores are calculated using the WHO growth standards. WAZ is used a proxy indicator of recent diarrhoea.
lost days at school and work | 21 months
healthcare expenditure | 21 months
latrine coverage and use | 21 months
bacteriological water quality | 21 months
fly counts | 21 months
Height-for-age | baseline and endline
  Recumbent length measured for children <2 at baseline and endline following standardised procedures for anthropometric assessment.
Diarrhoea (all ages) | 21 months
  Longitudinal prevalence of diarrhoea (7-day period prevalence) measured repeatedly every 3 months over a 21-month follow-up period. Diarrhoea is defined according to the WHO definition (passage of three or more loose stools in 24 hrs).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clasen, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Xavier Institute of Management, Bhubaneswar, Odisha, India

REFERENCES:
- [Derived] Routray P, Torondel B, Jenkins MW, Clasen T, Schmidt WP. Processes and challenges of community mobilisation for latrine promotion under Nirmal Bharat Abhiyan in rural Odisha, India. BMC Public Health. 2017 May 16;17(1):453. doi: 10.1186/s12889-017-4382-9. PMID 28511653
- [Derived] Freeman MC, Majorin F, Boisson S, Routray P, Torondel B, Clasen T. The impact of a rural sanitation programme on safe disposal of child faeces: a cluster randomised trial in Odisha, India. Trans R Soc Trop Med Hyg. 2016 Jul;110(7):386-92. doi: 10.1093/trstmh/trw043. PMID 27496512
- [Derived] Clasen T, Boisson S, Routray P, Torondel B, Bell M, Cumming O, Ensink J, Freeman M, Jenkins M, Odagiri M, Ray S, Sinha A, Suar M, Schmidt WP. Effectiveness of a rural sanitation programme on diarrhoea, soil-transmitted helminth infection, and child malnutrition in Odisha, India: a cluster-randomised trial. Lancet Glob Health. 2014 Nov;2(11):e645-53. doi: 10.1016/S2214-109X(14)70307-9. Epub 2014 Oct 9. PMID 25442689
- [Derived] Boisson S, Sosai P, Ray S, Routray P, Torondel B, Schmidt WP, Bhanja B, Clasen T. Promoting latrine construction and use in rural villages practicing open defecation: process evaluation in connection with a randomised controlled trial in Orissa, India. BMC Res Notes. 2014 Aug 1;7:486. doi: 10.1186/1756-0500-7-486. PMID 25084699